CLINICAL TRIAL: NCT02077777
Title: Azione Chemiopreventiva Della Mesalazina Sul Cancro Del Colon-retto: Studio Pilota Per la Valutazione Degli Effetti Molecolari "in Vivo" Sulla Via di Segnalazione Proliferativa Della β-catenina (Official Title in Italian Language)
Brief Title: Chemopreventive Action of Mesalazine on Colorectal Cancer: a Pilot Study for an "in Vivo" Evaluation of the Molecular Effects on β-catenin Signaling Pathway.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SOFAR S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MES-CT 01
Record Dates: First submitted 2014-02-28; First posted 2014-03-04 (Estimated); Last update posted 2016-12-02 (Estimated); Status verified 2016-12

CONDITIONS: Colorectal Cancer
Keywords: mesalazine; colon; cancer
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasms | interventions — Mesalamine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 5-ASA (Experimental): Mesalazine 800 mg orally t.i.d for 3 months
  Interventions: Drug: Mesalazine
- No treatment (No Intervention): no treatment

INTERVENTIONS:
Drug: Mesalazine — Mesalazine cpr 800 mg t.i.d. for 3 months
  Other Names: 5-aminosalicylic acid; 5-ASA; Pentacol
  Arms: 5-ASA

SUMMARY:
The purpose of this study is to obtain an "in vivo" confirmation that mesalazine induces the gene expression of μ-protocadherin and other related genes in the colon mucosa, as demonstrated in some "in vitro" experiments. .

DETAILED DESCRIPTION:
Pilot Trial, single-blind, parallel group on biopsy specimens of healthy colon mucosa in patients with precancerous lesions of the colon and rectum (adenomas) treated with mesalazine.

ELIGIBILITY:
Inclusion Criteria:

* Patients with precancerous colorectal lesions (polypoid or nonpolypoid adenomas) that needs of an endoscopic exam of control after 3 months from the removal of the lesions (determined on the basis of the morphological and histological characteristics of the lesions and of the removal technique)
* Ability and willingness to adhere to study regimen
* Written informed consent

The following inclusion criteria was deleted according to Amendment n. 01 approved by the Ethical Committee on 19/dec/2014:

- diverticular disease/diverticular colitis;

The rationale of this change is that the presence of diverticular disease/diverticular colitis does not contribute to the definition of the trial primary end-points and represents a critical point during the patient selection with an impact on duration and conduction of the study.

Exclusion Criteria:

* Patients under therapy with Aspirin (>100 mg/die) or other FANS
* Inflammatory bowel disease (IBD)
* Hypersensitivity to Mesalazine.
* Pregnant or nursing (lactating) women
* Patients who belonging to the category n. 4 of the ASA physical status classification system
* contraindications to mesalazine therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2012-10; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Molecular analysis of gene expression levels of μ-protocadherin and other related proteins | 3 months
  Molecular analysis (quantitative RT-PCR) of gene expression levels of μ-protocadherin, protocadherin 19, protocadherin 24, cadherin E, TCF7L2, TCF4, c-myc, Cyclin D1, p21waf1, VEGF, CD44, Met, KLF4 e CEBP-α and comparison of the levels assessed at the end of the treatment period with the baseline.

SECONDARY OUTCOMES:
Evaluation of protein expression level of μ-protocadherin, Ki-67, Caspase-3 and Histone H2AXγ, evaluation of DNA oxidative damage and intra-mucosal concentration of 5-Acetylsalicylic acid | 3 months
  These parameters will be examined using molecular analysis of the oxidation and depurination levels of the DNA and chromatographic analysis of the intra-mucosal concentration of 5-Acetylsalicylic acid, in biopsies of normal mucosa of the colon taken before and after the treatment of patients with 5-Acetylsalicylic acid:
  * quantification of the percentage of cells expressing the following proteins by immunohistochemical analysis: μ-protocadherin, Ki-67, Caspase-3 and Histone H2AXγ;
  * quantification of number of AP sites per 100000 DNA bp
  * quantification of nanograms di 8-OhdG (8-hydroxyguanine) per micrograms of DNA

CONTACTS AND LOCATIONS:
Overall Officials: Federico Buffoli, Doctor, Principal Investigator — Istituti Ospitalieri di Cremona
Locations (1):
- Istituti Ospitalieri di Cremona, Cremona, Cremona, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Parenti S, Ferrarini F, Zini R, Montanari M, Losi L, Canovi B, Ferrari S, Grande A. Mesalazine inhibits the beta-catenin signalling pathway acting through the upregulation of mu-protocadherin gene in colo-rectal cancer cells. Aliment Pharmacol Ther. 2010 Jan;31(1):108-19. doi: 10.1111/j.1365-2036.2009.04149.x. PMID 19785626
- [Background] Losi L, Parenti S, Ferrarini F, Rivasi F, Gavioli M, Natalini G, Ferrari S, Grande A. Down-regulation of mu-protocadherin expression is a common event in colorectal carcinogenesis. Hum Pathol. 2011 Jul;42(7):960-71. doi: 10.1016/j.humpath.2010.10.009. Epub 2011 Mar 2. PMID 21315419
- [Background] Brown JB, Lee G, Managlia E, Grimm GR, Dirisina R, Goretsky T, Cheresh P, Blatner NR, Khazaie K, Yang GY, Li L, Barrett TA. Mesalamine inhibits epithelial beta-catenin activation in chronic ulcerative colitis. Gastroenterology. 2010 Feb;138(2):595-605, 605.e1-3. doi: 10.1053/j.gastro.2009.10.038. Epub 2009 Oct 29. PMID 19879273
- [Background] Velayos FS, Terdiman JP, Walsh JM. Effect of 5-aminosalicylate use on colorectal cancer and dysplasia risk: a systematic review and metaanalysis of observational studies. Am J Gastroenterol. 2005 Jun;100(6):1345-53. doi: 10.1111/j.1572-0241.2005.41442.x. PMID 15929768
- [Background] Lyakhovich A, Gasche C. Systematic review: molecular chemoprevention of colorectal malignancy by mesalazine. Aliment Pharmacol Ther. 2010 Jan 15;31(2):202-9. doi: 10.1111/j.1365-2036.2009.04195.x. Epub 2009 Nov 5. PMID 19891667
- [Background] Gushima M, Hirahashi M, Matsumoto T, Fujita K, Fujisawa R, Mizumoto K, Nakabeppu Y, Iida M, Yao T, Tsuneyoshi M. Altered expression of MUTYH and an increase in 8-hydroxydeoxyguanosine are early events in ulcerative colitis-associated carcinogenesis. J Pathol. 2009 Sep;219(1):77-86. doi: 10.1002/path.2570. PMID 19479711
- [Background] Obtulowicz T, Swoboda M, Speina E, Gackowski D, Rozalski R, Siomek A, Janik J, Janowska B, Ciesla JM, Jawien A, Banaszkiewicz Z, Guz J, Dziaman T, Szpila A, Olinski R, Tudek B. Oxidative stress and 8-oxoguanine repair are enhanced in colon adenoma and carcinoma patients. Mutagenesis. 2010 Sep;25(5):463-71. doi: 10.1093/mutage/geq028. Epub 2010 Jun 9. PMID 20534734